CLINICAL TRIAL: NCT04520438
Title: Effect of Leucocyte and Platelet Rich Fibrin as an Adjuvant in Non-Surgical Periodontal Therapy: A Split-Mouth Randomized Controlled Clinical Trial
Brief Title: L-PRF Plus Non Surgical Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Responsible Party: Principal Investigator, Catherine Andrade, Principal investigator, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSPT + L-PRF
Record Dates: First submitted 2020-08-12; First posted 2020-08-20 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Periodontitis
Keywords: Platelet-Rich Fibrin; Chronic Chronic Periodontitis; Dental Scaling; Root Planing; Gingival Crevicular Fluid; Microbiology
MeSH Terms: conditions — Periodontitis; Chronic Periodontitis | interventions — Leukocyte Count; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: A split-mouth, randomized controlled clinical trial enrolling 13 patients (8 males and 5 females, mean age 52.3 ± 9.4 years) was set-up. The periodontal pockets ≥ 6 mm were randomly treated with SRP + L-PRF (test group) or SRP alone (control group)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Only the clinician who provided the treatment knew the treatment assigned. A different clinician performed all the evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NSPT + L-PRF (Experimental): Scaling and root planing associated to Leucocyte and Platelet rich Fibrin Membrane and irrigation with exudate of L-PRF.
  Interventions: Procedure: Leukocyte and platelet rich fibrin; Procedure: Non-Surgical Periodontal treatment
- NSPT alone (Other): Only Scaling and root planing
  Interventions: Procedure: Non-Surgical Periodontal treatment

INTERVENTIONS:
Procedure: Leukocyte and platelet rich fibrin — L-PRF membrane and irrigation with L-PRF exudate in the same treatment session of NSPT
  Other Names: L-PRF
  Arms: NSPT + L-PRF
Procedure: Non-Surgical Periodontal treatment — The control group only received NSPT (scaling and root planing) in one treatment session.
  Other Names: Scaling and root planing

SUMMARY:
Abstract:

Background: Leucocyte and Platelet-Rich Fibrin (L-PRF) has shown to promote regenerative processes, even reporting antibacterial effect. The aim of this split-mouth clinical trial was to evaluate the effect of L-PRF as an adjuvant to scaling and root planing (SRP).

Methods: 13 patients with chronic periodontitis and at least 1 bilateral periodontal pocket ≥ 6 mm were recruited. The sites were randomly treated with SRP + L-PRF (test group) or SRP alone (control group). The following parameters were evaluated at baseline and 6 weeks, 3 and 6 months after treatment: Probing pocket depth (PPD), clinical attachment level (CAL), bleeding on probing (BOP); gingival recession (GR), and root sensitivity (RS). Additionally, the concentrations of Porphyromona gingivalis (P.g), Aggregatibacter actinomycetemcomitans (A.a), Prevotella intermedia (P.i) and Fusobacterium nucleatum (F.n) in the gingival crevicular fluid (GCF) were evaluated at baseline, 6 weeks and 3 months after treatment.

DETAILED DESCRIPTION:
Materials and Methods Study design and Patient Selection A split-mouth, randomized controlled clinical trial enrolling 13 patients (8 males and 5 females, mean age 52.3 ± 9.4 years) was set-up. The patients were informed about the benefits and risks of the study and each participant signed informed consent.

Non-surgical periodontal treatment A single periodontist (L.C.) performed all periodontal treatments. NSPT consisted of two sessions of scaling and root planing (SRP) within 48 hours under local anesthesia using ultrasonic and hand instrumentation. Additionally, the sites associated with PPD ≥ 6 mm in the quadrant assigned to the test group were irrigated with L-PRF exudate and filled with longitudinal pieces of L-PRF membrane. The patients received instructions about soft diet, a carefully and soft mouth rinse with chlorhexidine 0.12%, and no toothbrushing during 7 days in order to avoid the L-PRF removal. After this period, the following instructions were given: modified Bass brushing technique, dental floss, and interdental brushes, and chlorhexidine 0.12% mouth rinse for an extra 7 days. Strict hygiene control by the clinician was also performed in each appointment.

L-PRF membrane preparation Two samples of venous blood were collected in 2 vacutainer tubes (red cup) of 10 ml without anticoagulant. They were centrifuged at 408 g for 12 minutes using a table centrifuge (IntraSpinTM, Intralock®, Florida, USA) according to the protocol described by Temmerman et al.18 The L-PRF clots were removed from the tube, separated from the red cells and placed in the Xpression box (IntraSpinTM, Intralock®, Florida, USA) to gently compress them in membranes. The membranes were chopped in longitudinal pieces to fill the periodontal pockets ≥ 6mm. The exudate, released during the compression, called L-PRF exudate was aspirated to rinse the treated pockets. (Figure 1)

Clinical Measurements All clinical measurements were performed by a single trained and calibrated examiner (N.J.) who was masked for the treatment assigned, using a basic examination instrument kit and a University of North Carolina no. 15 color-coded periodontal probe. The following clinical parameters were measured at baseline and 6 weeks, 3 months and 6 months after treatment: probing pocket depth (PPD), clinical attachment level (CAL), gingival recession (GR), bleeding on probing (BOP), and O´Leary plaque index (PI).19 Additionally, the root sensitivity (RS) was evaluated using a 100-mm visual analogue scale (VAS) (0 indicating no pain, 50 indicating average, and 100 indicating an unbearable pain) at 24 hrs., 6 weeks, 3 months, and 6 months after treatment. The change in PPD, CAL, GR, BOP, PI, and RS (difference between baseline measures and at 1, 3, and 6 months) were calculated.

GCF collection GCF samples were collected from the deepest pocket from each quadrant before recording the clinical measurement (baseline, and 6 weeks and, 3 months after treatment) in order to evaluate the concentration of Porphyromona gingivalis (P.g), Aggregatibacter actinomycetemcomitans (A.a), Prevotella intermedia (P.i) and Fusobacterium nucleatum (F.n). The sample area was isolated with cotton rolls, and contamination with saliva was avoided using an appropriate suction and air spray. Then, an endodontic #35 paper-point was inserted until a slight resistance was felt and it was held for 30 seconds. The paper-points were immediately inserted in an Eppendorf tube and stored at -80ºC for future analysis.

Microbiological processing After defrosting the samples, 1ml of phosphate-buffered saline (PBS) was added and homogenized. Then, 400 μl of each sample was centrifuged at 13200 rpm for 3 minutes. The obtained pellet was dispersed in 200 μl InstaGene. DNA was extracted with InstaGene matrix (Bio-Rad Life Science Research, Hercules, CA, USA) according to the instructions of the manufacturer. Five microliters of the purified DNA were used for the quantification of Porphyromonas gingivalis, Aggregatibacter actinomycetemcomitans, Fusobacterium nucleatum, and Prevotella intermedia. A quantitative polymerase chain reaction (qPCR) assay was performed with a CFX96 Real-Time System (Biorad, Hercules, CA, USA) using the Taqman 5' nuclease assay PCR method for detection and quantification of bacterial DNA. Taqman reaction contained 12.5 μl Mastermix (Eurogentec, Seraing, Belgium), 4.5 μl sterile distilled water, 1 μl of both species-specific primers and probe (Table 1) and 5 μl template DNA. Assay conditions for all primer/probe set consisted of an initial 2 min at 50°C, followed by a denaturation step for 10 min at 95°C, followed by 45 cycles of 95°C for 15 sec and 60°C for 60 sec. Quantification was based on a plasmid standard curve. The delta for bacterial concentration at 6 weeks, 3 and 6 months (difference between baseline measures and at 6 weeks, 3 and 6 months) were calculated.

Randomization, allocation concealment and calibration A coin toss method was used to assign the patients' quadrants into two treatment groups: (SRP + L-PRF) or control (SRP alone).

Before beginning the study, two recordings of the following parameters were done: PPD, GR, and CAL in five patients, with a 24-hour interval between first and second records in order to validate the intra-examiner accuracy. All teeth, excluding third molars, were measured by periodontal probing at 6 sites (mesiobuccal, mediobuccal, distobuccal, mesiolingual/palatal, mediolingual/palatal, and distolingual/palatal). Calibration was accepted if the measurements at baseline and after 24 hours were within 1 mm at the 95% level (correlation coefficients between duplicate measurements; r = 0.95).

Statistical analysis To detect a mean difference in PPD of 1.2 mm with a standard deviation of 1.0 at an α level of 0.05 and a β level of 0.10 (power = 0.9), a sample size of 10 patients was required. Despite the results but to anticipate potential drop outs during the study, a sample size of n = 16 patients was considered.

Bacterial counts were log-transformed. A linear mixed model was applied with the variable patient, as a random factor and time and treatment as two crossed fixed factors. Smoking and PI were considered as covariables. Contrasts were set up to calculated the change from baseline for the different time points between the treatments and for each treatment apart. A correction for simultaneous hypothesis testing according to Sidak was applied. A normal quantile plot and residual dot plot of the residual values were created showing that the assumptions underlying the statistical model could be made.

ELIGIBILITY:
Inclusion Criteria:

* age between 30 and 70 years old
* diagnosis of chronic periodontitis
* at least one bilateral periodontal pocket ≥ 6 mm
* healthy patients

Exclusion Criteria:

* inability to comply with the study protocol
* receiving antibiotic therapy or non-steroidal anti-inflammatory drugs during the previous two months or using calcium channel blockers, phenytoin, cyclosporine, or any associated drug that might affect gingival tissue
* periodontal treatment during the previous 12 months
* auto-immune disorders (self-reported)
* requiring antibiotic prophylaxis before periodontal treatment; or requiring non-steroidal anti-inflammatory drugs for postoperative pain management after periodontal treatment
* smokers >10 cigarettes
* pregnancy/lactation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline pocket probing depth at 6 weeks | 6 weeks
  Change from baseline to 6 weeks of the distance from the gingival margin to the base of the clinical pocket for each site. Unit: millimeters
Change from baseline pocket probing depth at 3 months | 3 months
  Change from baseline to 3 months of the distance from the gingival margin to the base of the clinical pocket for each site. Unit: millimeters
Change from baseline pocket probing depth at 6 months | 6 months
  Change from baseline to 6 months of the distance from the gingival margin to the base of the clinical pocket for each site. Unit: millimeters

SECONDARY OUTCOMES:
Change from baseline clinical attachment level at 6 weeks | 6 weeks
  Change from baseline to 6 weeks of the distance between the base of the clinical pocket and the cement-enamel junction. Unit: millimeters
Change from baseline clinical attachment level at 3 months | 3 months
  Change from baseline to 3 months of the distance between the base of the clinical pocket and the cement-enamel junction. Unit: millimeters
Change from baseline clinical attachment level at 6 months | 6 months
  Change from baseline to 6 months of the distance between the base of the clinical pocket and the cement-enamel junction. Unit: millimeters
Change from baseline gingival recession at 6 weeks | 6 weeks
  Change from baseline to 6 weeks of the distance between gingival margin and the cement-enamel junction. Unit: millimeters
Change from baseline gingival recession at 3 months | 3 months
  Change from baseline to 3 months of the distance between gingival margin and the cement-enamel junction. Unit: millimeters
Change from baseline gingival recession at 6 months | 6 months
  Change from baseline to 6 months of the distance between gingival margin and the cement-enamel junction. Unit: millimeters
Change from baseline bleeding on probing at 6 weeks | 6 weeks
  Change from baseline to 6 weeks of the percentage of sites with bleeding on probing
Change from baseline bleeding on probing at 3 months | 3 months
  Change from baseline to 3 months of the percentage of sites with bleeding on probing
Change from baseline bleeding on probing at 6 months | 6 months
  Change from baseline to 6 months of the percentage of sites with bleeding on probing
Change from baseline O´Leary plaque index at 6 weeks | 6 weeks
  Change from baseline to 6 weeks of percentage of surfaces with dental plaque (100% to 0%)
Change from baseline O´Leary plaque index at 3 months | 3 months
  Change from baseline to 3 months of percentage of surfaces with dental plaque (100% to 0%)
Change from baseline O´Leary plaque index at 6 months | 6 months
  Change from baseline to 6 months of percentage of surfaces with dental plaque (100% to 0%)
Change from baseline root sensitivity at 24 hours | 24 hours
  Change from baseline to 24 hours of Intensity of root sensitivity according to visual analogue scale (0 indicating no pain, 50 indicating average, and 100 indicating an unbearable pain)
Change from baseline root sensitivity at 6 weeks | 6 weeks
  Change from baseline to 6 weeks of Intensity of root sensitivity according to visual analogue scale (0 indicating no pain, 50 indicating average, and 100 indicating an unbearable pain)
Change from baseline root sensitivity at 3 months | 3 months
  Change from baseline to 3 months of Intensity of root sensitivity according to visual analogue scale (0 indicating no pain, 50 indicating average, and 100 indicating an unbearable pain)
Change from baseline root sensitivity at 6 months | 6 months
  Change from baseline to 6 months of Intensity of root sensitivity according to visual analogue scale (0 indicating no pain, 50 indicating average, and 100 indicating an unbearable pain)
Change from baseline microbiological assessment in gingival crevicular fluid at 6 weeks | 6 weeks
  Change from baseline to 6 weeks of quantification of Porphyromonas gingivalis, Aggregatibacter actinomycetemcomitans, Fusobacterium nucleatum and Prevotella intermedia by quatitative polymerase chain reaction
Change from baseline microbiological assessment in gingival crevicular fluid at 3 months | 3 months
  Change from baseline to 3 months of quantification of Porphyromonas gingivalis, Aggregatibacter actinomycetemcomitans, Fusobacterium nucleatum and Prevotella intermedia by quatitative polymerase chain reaction

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Andrade, DDs, Principal Investigator — Universidad de Los Andes
Locations (1):
- Universidad de Los Andes, Santiago, Chile